CLINICAL TRIAL: NCT04823780
Title: Investigation of the Effects of Early Enteral Nutrition on Endoscopic Therapy of Esophagogastric Varices in Liver Cirrhosis:An Observational Study
Brief Title: The Effects of Early Enteral Nutrition on Endoscopic Therapy of Esophagogastric Varices in Liver Cirrhosis
Status: Completed | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: 20200901-Qilu
Record Dates: First submitted 2021-02-04; First posted 2021-04-01 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2021-03

CONDITIONS: Liver Cirrhosis; Esophageal and Gastric Varices
Keywords: Early enteral nutrition; Esophageal and Gastric Varices; Rebleeding
MeSH Terms: conditions — Liver Cirrhosis; Esophageal and Gastric Varices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- early enteral nutrition support group: Nutrient solution is provided through oral nutrient solution within 4-48 hours after endoscopic treatment
  Interventions: Dietary Supplement: nutrient solution
- parenteral Nutrition Group: Intravenous nutrition is provided within 48 hours after endoscopic treatment

INTERVENTIONS:
Dietary Supplement: nutrient solution — For the patients with esophageal and gastric varices after endoscopic treatment，start taking the nutrient solution at the fourth hour.
  Groups: early enteral nutrition support group

SUMMARY:
The purpose of this study was to evaluate the safety of early enteral nutrition on endoscopic therapy of esophagogastric varices in Liver Cirrhosis ,and to assess the impact of different eating times on patients, so as to determine the best time for patients to obtain nutrition after surgery.

DETAILED DESCRIPTION:
For patients with gastroesophageal varices in Liver Cirrhosis,, there is no clear guideline and consensus on when to start eating after endoscopic treatment. In 2015, a randomized controlled study in Taiwan of China confirmed that compared with liquid diet given 48 h after endoscopic treatment, liquid diet given 4 h and started enteral nutrition would not increase the risk of rebleeding, and could improve the nutritional status of patients. However, some patients after endoscopic treatment would suffer from post-sternal pain, abdominal pain, nausea, vomiting and other discomforts, affecting appetite and delay the diet time. Based on the above research background, we observed and evaluated the safety and effectiveness of early enteral nutrition in patients with cirrhotic esophageal and gastric varices after endoscopic treatment, and analyzed the influencing factors of enteral nutrition in patients with cirrhotic esophageal and gastric varices after endoscopic treatment, so as to further clarify the optimal time for patients to eat after endoscopic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cirrhosis of gastroesophageal varices undergoing endoscopic therapy

Exclusion Criteria:

* Endoscopic treatment of uncontrollable bleeding
* Accompanied with other endoscopic treatments that need to be fasting
* With obvious hepatic encephalopathy and liver failure
* Did not sign the informed consent form and refused to participate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cirrhosis of gastroesophageal varices undergoing endoscopic
Sampling Method: Non-Probability Sample
Enrollment: 397 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-10-20 (Actual)

PRIMARY OUTCOMES:
rebleeding | 2 to 30days
  the rate of rebleeding after endoscopic therapy

CONTACTS AND LOCATIONS:
Overall Officials: Gao Yanjing, PhD.MD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital , Shandong University, Jinan, Shandong, China

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-01): https://cdn.clinicaltrials.gov/large-docs/80/NCT04823780/Prot_SAP_000.pdf